CLINICAL TRIAL: NCT04286295
Title: Pilot RCT of Cytisine Compared to Combination Nicotine Replacement Therapy to Reduce Cigarette Consumption in Relapsed Smokers
Brief Title: Cytisine Compared to Combination NRT in Relapsed Smokers
Acronym: CYTvsNRT+
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190720-01H
Record Dates: First submitted 2020-02-21; First posted 2020-02-26 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Smoking Cessation; Coronary Artery Disease
Keywords: Tobacco; Relapse prevention
MeSH Terms: conditions — Smoking Cessation; Coronary Artery Disease | interventions — cytisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cytisine (Experimental): Cravv™ (Zpharm, Waterloo) is a natural health product licensed by Health Canada to assist with smoking cessation; each oral capsule contains 1.5mg of cytisine. The dosing is as follows: 6 capsules daily for the first 3 days; 5 capsules daily for days 4-12; 4 capsules daily for days 13-16; 3 capsules daily for days 17-20; and 1-2 capsules daily for days 21-25.
  Interventions: Drug: Cytisine
- NRT+ (Active Comparator): The Nicoderm® patch plus Nicorette® Lozenge will be provided to participants in the combination NRT group. Participants smoking less than 15 cigarettes per day will be provided with 14 mg patches while those smoking 15 or more cigarettes per day will receive 21 mg patches. Participants will be told to apply a new patch each morning. Participants will be instructed to use the lozenges as needed (up to 15 per day) to overcome nicotine cravings. Lozenges are available in both 2mg and 4mg strengths. For those who are smoking less than 15 cigarettes per day, they will be given the 2mg strength. For those who are smoking 15 or more cigarettes per day, they will receive the 4mg strength.
  Interventions: Drug: Nicoderm C-Q Transdermal Product; Drug: Nicorette Lozenge Product

INTERVENTIONS:
Drug: Cytisine — Cytisine is a plant-based smoking cessation medication. Cytisine acts by reducing the rewarding effect of nicotine and attenuating nicotine withdrawal symptoms. A recent review concluded that cytisine is the most promising future smoking cessation treatment. Cytisine is inexpensive to produce and is currently priced much lower than other cessation medications. It is well-tolerated by smokers and requires a shorter treatment period than conventional treatments. Because it is plant-based, cytisine may be attractive for smokers who prefer 'natural' medicines. Numerous placebo-controlled studies have demonstrated the safety and efficacy of cytisine. One high-quality pragmatic non-inferiority trial (n = 1310) found that cytisine was superior to nicotine replacement therapy (NRT) in improving self-reported continuous abstinence rates at 1 week, and 1, 2 and 6 months when both groups received minimal behavioural support.
  Arms: Cytisine
Drug: Nicoderm C-Q Transdermal Product — The Nicoderm® patch plus Nicorette® Lozenge will be provided to participants in the combination NRT group. Participants will be instructed to apply a new patch each day. They will continue to wear patches for 25 days.
  Other Names: NRT+
  Arms: NRT+
Drug: Nicorette Lozenge Product — Participants in the NRT group will receive Nicorette Lozenges to use during their 25-day quit attempt. They will receive enough lozenges to last for the 25-day treatment period.
  Arms: NRT+

SUMMARY:
Cigarette smoking causes cardiovascular disease (CVD) yet many smokers with CVD are unable to quit despite strong desire to do so. Within 90 days of discharge, about 30% of smokers have returned to daily smoking and almost 60% have relapsed by 1 year. Patients with CVD who resume smoking are more likely to experience new events (e.g. heart attack or stroke) or die. New approaches are required. A new type of cessation product is a plant-based medication called Cytisine. Cytisine is taken orally over 25 days and reduces the pleasurable sensations that smokers get from cigarettes and reduces withdrawal symptoms. The primary research question is whether or not it is feasible to conduct a large-scale trial of the effectiveness of this product compared to conventional nicotine replacement therapy in smokers who have failed to quit using conventional methods. To determine feasibility, a pilot study will be conducted of sixty smokers (30 men, 30 women) with CVD who have been treated for smoking cessation but have relapsed within 90 days of discharge. Participants will complete a baseline assessment and will be randomly assigned to either the combination nicotine replacement therapy group (patch plus lozenge) or cytisine group. Participants will be treated for 25 days and then will return to UOHI so adherence to treatment and smoking status can be assessed. Feasibility of the larger trial will be based on: the recruitment rates; adherence to assigned treatments; dropout rates; and differences in 25-day quit rates between groups.

DETAILED DESCRIPTION:
Cigarette smoking is a causative factor in the development of coronary heart disease (CHD), and is the most dangerous form of tobacco use. Effective treatments for smoking cessation exist but relapse to cigarette smoking is common, principally due to nicotine addiction and related symptoms of withdrawal. Little is known about how best to support smokers who have relapsed in subsequent attempts to change their smoking behavior. One emerging treatment has features that might make it appealing to smokers and may be effective in the setting of recent relapse: cytisine.

Cytisine is a plant-based smoking cessation medication with more than 50 years of use in central/eastern Europe. Cytisine is a partial agonist of nicotinic acetylcholine receptors (nAChRs), which is central to the effect of nicotine on the reward pathway. Cytisine acts by reducing the rewarding effect of nicotine and attenuating nicotine withdrawal symptoms. A recent review concluded that cytisine is the most promising future smoking cessation treatment. Cytisine is inexpensive to produce and is currently priced much lower than other cessation medications. It is well-tolerated by smokers and requires a shorter treatment period (i.e. 25 days) than conventional treatments. Because it is plant-based, cytisine may be attractive for smokers who prefer 'natural' medicines. Numerous placebo-controlled studies have demonstrated the safety and efficacy of cytisine. One high-quality pragmatic non-inferiority trial (n = 1310) found that cytisine was superior to nicotine replacement therapy (NRT) in improving self-reported continuous abstinence rates at 1 week, and 1, 2 and 6 months when both groups received minimal behavioural support. In Canada, cytisine is marketed as the natural health product Cravv™.

The long-term goal is to conduct a definitive, large-scale randomized controlled trial (RCT) of the efficacy of cytisine compared to conventional treatment (i.e. combination NRT) for smoking cessation among smokers who have relapsed to smoking following hospitalization for a CHD-related event. Prior to conducting a larger, definitive RCT there is a need to conduct a pilot study to better understand the potential feasibility of such a trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is enrolled in UOHI's Quit Smoking Program;
2. Patient has relapsed to daily smoking ≥10 cigarettes per day within 90 days of discharge from UOHI;
3. Patient is currently smoking ≥10 cigarettes per day.

Exclusion Criteria:

1. Patient has used NRT, cytisine, varenicline, bupropion or a nicotine-containing vaping device within in the past 15 days;
2. Patient is unavailable to come to UOHI for assessments;
3. Patient is unable to provide informed consent;
4. Patient is unable to comprehend the intervention instructions (in the opinion of qualified investigators)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of study | Baseline to 25-day follow-up
  will be feasible to recruit 10 relapsed smokers with CHD per month to a study of cytisine vs. combination NRT

SECONDARY OUTCOMES:
Treatment completion | Baseline to 25-day follow-up
  Participants will complete at least 70% of their prescribed treatment
Attrition | Baseline to 25-day follow-up
  There will be less than 5% attrition over a 25-d treatment period
Cigarette consumption | Baseline to 25-day follow-up
  Cigarette consumption will drop by 5 cigs/d more in the cytisine group compared to the combination NRT group by the end of the 25-d treatment period
Arterial Stiffness | Baseline to 25-day follow-up
  Arterial stiffness, as measured by pulse wave velocity, will improve in smokers who are able to achieve complete abstinence (i.e. smoking zero cigarettes per day).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pipe, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Insitute - Prevention and Wellness Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This is a pilot study so datasets will not be shared until a written request is submitted to the PI.

REFERENCES:
- [Derived] Mir H, Mullen KA, Heshmati J, Baldwin A, Quirouette E, Serano E, Coja M, Pipe AL, Reid RD. Cytisine Use Vs Nicotine Replacement Therapy in Relapsed Smokers with Heart Disease: Feasibility Results from a Pilot Randomized Trial. CJC Open. 2025 May 16;7(8):1062-1069. doi: 10.1016/j.cjco.2025.05.005. eCollection 2025 Aug. PMID 40894854
- [Derived] Mir H, Heshmati J, Mullen KA, Baldwin A, Quirouette E, Pipe A, Reid R. Cytisine compared to combination nicotine replacement therapy to reduce cigarette consumption in relapsed smokers: protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2025 Jan 28;11(1):10. doi: 10.1186/s40814-024-01591-4. PMID 39876021